CLINICAL TRIAL: NCT07265804
Title: Current Regenerative Approaches Applied to Immature Teeth With Necrotic Pulps
Brief Title: PRF and CGF Scaffolds With EDTA in Regeneration
Acronym: RET-EDTA-CGF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Aliye Kamalak, Assoc. Prof., Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RET-EDTA-Study-2024; 2024/3-14 D (Other Grant/Funding Number: Scientific Research Projects Unit of KSU,Turkey)
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pulp Necrosis; Immature Permanent Teeth; Open Apex; Periapical Periodontitis; Procedure
Keywords: Regenerative Endodontics; Platelet-Rich Fibrin; Concentrated Growth Factor; Blood Clot Scaffold; EDTA Irrigation
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis | interventions — Blood Coagulation; Edetic Acid; Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group interventional model in which 30 immature permanent teeth diagnosed with pulp necrosis were randomly assigned to six treatment arms. Each participant received only one intervention, consisting of one scaffold type (blood clot, PRF, or CGF) combined with either 5% or 17% EDTA as the final irrigant. All groups were treated and followed simultaneously, and no crossover occurred between interventions.
Masking Description: No blinding was possible because the type of scaffold (blood clot, PRF, or CGF) and the EDTA concentration (5% or 17%) were visibly identifiable during the clinical procedure. Operators could not be masked, and participants were aware of the treatment steps, making the study open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Blood Clot + 5% EDTA (Experimental): Standard regenerative endodontic treatment using final irrigation with 5% EDTA followed by induction of bleeding to form a blood clot scaffold.
  Interventions: Procedure: Blood Clot + 5% EDTA
- Blood Clot + 17% EDTA (Experimental): Regenerative endodontic procedure using final irrigation with 17% EDTA and blood clot scaffold formation.
  Interventions: Procedure: Blood Clot + 17% EDTA
- PRF + 5% EDTA (Experimental): Regenerative endodontic procedure using platelet-rich fibrin scaffold after final irrigation with 5% EDTA.
  Interventions: Procedure: PRF + 5% EDTA
- PRF + 17% EDTA (Experimental): Regenerative endodontic procedure using platelet-rich fibrin scaffold following final irrigation with 17% EDTA.
  Interventions: Procedure: PRF + 17% EDTA
- CGF + 5% EDTA (Experimental): Regenerative endodontic protocol using concentrated growth factor scaffold after final irrigation with 5% EDTA.
  Interventions: Procedure: CGF + 5% EDTA
- CGF + 17% EDTA (Experimental): Regenerative endodontic procedure using concentrated growth factor scaffold following final irrigation with 17% EDTA.
  Interventions: Procedure: CGF + 17% EDTA

INTERVENTIONS:
Procedure: Blood Clot + 5% EDTA — Final irrigation with 5% EDTA followed by induction of apical bleeding to form an intracanal blood clot scaffold as part of the regenerative endodontic procedure.
  Arms: Blood Clot + 5% EDTA
Procedure: Blood Clot + 17% EDTA — Final irrigation with 17% EDTA followed by controlled induction of bleeding beyond the apex to produce a blood clot scaffold for regenerative endodontic treatment.
  Arms: Blood Clot + 17% EDTA
Procedure: PRF + 5% EDTA — Application of platelet-rich fibrin (PRF) scaffold after final irrigation with 5% EDTA during regenerative endodontic therapy.
  Arms: PRF + 5% EDTA
Procedure: PRF + 17% EDTA — Use of platelet-rich fibrin (PRF) scaffold following final irrigation with 17% EDTA in regenerative endodontic treatment.
  Arms: PRF + 17% EDTA
Procedure: CGF + 5% EDTA — Placement of concentrated growth factor (CGF) scaffold after final irrigation with 5% EDTA as part of the regenerative endodontic protocol.
  Arms: CGF + 5% EDTA
Procedure: CGF + 17% EDTA — Placement of concentrated growth factor (CGF) scaffold following final irrigation with 17% EDTA during regenerative endodontic treatment.
  Arms: CGF + 17% EDTA

SUMMARY:
This study evaluated the regenerative outcomes of immature permanent teeth with necrotic pulps treated using three scaffold types-blood clot, platelet-rich fibrin (PRF), and concentrated growth factor (CGF)-combined with either 5% or 17% EDTA as the final irrigant. Thirty teeth were randomly assigned to six treatment groups and followed clinically and radiographically for 12 months. Cone-beam computed tomography (CBCT) was used to assess root development parameters, including root length increase, apical diameter change, hard tissue formation, and periapical lesion volume. Clinical assessments included pain, swelling, sinus tract formation, percussion sensitivity, and pulp sensitivity testing. The study aimed to determine whether different scaffold materials and EDTA concentrations influence regenerative healing responses in immature necrotic teeth.

DETAILED DESCRIPTION:
This prospective randomized clinical study investigated regenerative endodontic treatment approaches for immature permanent teeth diagnosed with pulp necrosis and associated periapical pathology. Thirty teeth were allocated into six treatment subgroups based on two variables: scaffold type (blood clot, platelet-rich fibrin [PRF], or concentrated growth factor [CGF]) and final irrigation protocol (5% EDTA or 17% EDTA). All procedures were performed using a standardized regenerative protocol that included sodium hypochlorite irrigation, intracanal antibiotic medication, induction of apical bleeding when applicable, placement of the assigned scaffold, coronal sealing with mineral trioxide aggregate (MTA), and final composite restoration.

Radiographic evaluation involved cone-beam computed tomography (CBCT) at baseline and 12 months to measure root length development, apical diameter changes, hard tissue formation, and volumetric alterations in periapical lesions. Periapical radiographs were taken at baseline, 6 months, and 12 months to complement CBCT findings. Clinical follow-up included assessment of symptoms such as pain, swelling, sinus tract presence, tenderness to percussion, and pulp sensitivity using cold testing and electric pulp testing.

The primary aim of this study was to compare the effects of scaffold type and EDTA concentration on the biological and radiographic outcomes of regenerative endodontic treatment. The study sought to clarify how these variables may influence root maturation, apical closure, pulp vitality responses, and periapical tissue healing within a regenerative framework. This research was designed to contribute to the optimization of clinical protocols for managing immature teeth with necrotic pulps.

ELIGIBILITY:
Inclusion Criteria:

* Immature permanent teeth with open apices
* Diagnosis of pulp necrosis
* Radiographic evidence of periapical pathology
* Teeth suitable for isolation and restoration
* Patients aged 9 to 25 years
* No systemic diseases that contraindicate dental treatment
* Willingness to attend follow-up visits
* Signed informed consent by patient or guardian

Exclusion Criteria:

* Teeth with root fractures
* Teeth with severe canal curvature (>30°)
* Teeth with advanced root resorption
* Periodontal pocket depth >3 mm
* Previous endodontic treatment or retreatment
* Pregnancy
* Use of antibiotics or analgesics within the last 7 days
* Nonrestorable crowns
* Uncooperative patients unable to attend follow-up

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Root Length Increase | Baseline to 12 months
  Increase in root length measured using cone-beam computed tomography (CBCT).

SECONDARY OUTCOMES:
Apical Diameter Change (Apical Closure) | Baseline to 12 months
  Change in apical diameter measured by CBCT, used to evaluate apical closure after regenerative treatment.
Periapical Lesion Volume Reduction | Baseline to 12 months
  Volumetric reduction in periapical radiolucency measured by CBCT segmentation.
Hard Tissue Formation Volume | Baseline to 12 months
  Increase in newly formed mineralized tissue volume assessed by CBCT 3D segmentation.
Pulp Sensitivity Response | 12 months
  Presence or absence of a positive response to cold testing and electric pulp testing (EPT).
Clinical Healing | Baseline, 6 months, and 12 months
  Absence of pain, swelling, sinus tract, and percussion sensitivity during follow-up examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Aliye Kamalak, Principal Investigator — Kahramanmaraş Sütçü İmam University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Kahramanmaraş Sütçü İmam University, Faculty of Dentistry, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD), including CBCT images and clinical records, will not be shared due to patient confidentiality and ethical restrictions stated by the institutional review board.